CLINICAL TRIAL: NCT00087763
Title: A Phase II Prospective, Randomized, Double-Masked, Sham-Controlled, Dose-Ranging, Multi-Center Trial to Assess the Effect of Pegaptanib Sodium on Foveal Thickening in Patients With Exudative Subfoveal Age-Related Macular Degeneration (AMD)
Brief Title: Pegaptanib Sodium on Foveal Thickening in Patients With Exudative Subfoveal Age-Related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eyetech Pharmaceuticals (Industry)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: EOP 1009
Record Dates: First submitted 2004-07-13; First posted 2004-07-16 (Estimated); Last update posted 2006-05-03 (Estimated); Status verified 2006-05

CONDITIONS: Macular Degeneration
Keywords: AMD; Age Related Macular Degeneration; Exudative Subfoveal Age Related Macular Degeneration with Subfoveal Choroidal Neovascularization
MeSH Terms: conditions — Macular Degeneration | interventions — pegaptanib

INTERVENTIONS:
Drug: Macugen ™ (pegaptanib sodium injection)

SUMMARY:
The purpose of this study is to determine if Macugen™ reduces foveal thickness and improves vision in patients with wet AMD.

DETAILED DESCRIPTION:
This will be a randomized, double-masked, controlled, dose-ranging, multi-center comparative trial, in parallel groups. Patients will be stratified by clinical center and foveal thickness to be treated either Macugen or a sham injection. After 24 weeks, all patients will treated with Macugen until the end of the study at 54 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Best corrected visual acuity in the study eye between 20/40 and 20/320 and better or equal to 20/800 in the fellow eye.
* Foveal thickness <= 300 um (measured by OCT center point thickness).
* Subfoveal choroidal neovascularization secondary to age-related macular degeneration, with a total lesion size (including blood, scar/atrophy & neovascularization) of <= 12 disc areas, of which at least 50% must be active CNV.

Exclusion Criteria:

* Previous subfoveal thermal laser therapy.
* Any subfoveal atrophy or scarring, blood over the fovea, or fibrosis. Additionally no more than 25% of the total lesion size may be made up of scarring or atrophy.
* Previous photodynamic therapy with Visudyne (PDT) in the study eye. Eyes with predominantly classic lesions (as classified by fluorescein angiographic appearance) may be enrolled in the trial if, in the clinical judgment of the investigator, PDT can be deferred for at least 54 weeks after the first study treatment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135
Dates: Start 2004-03; Study Completion 2006-05